CLINICAL TRIAL: NCT00387439
Title: ORALIA Trial Randomized Controlled Trial of Medical Treatment Alone vs Medical Treatment Associated With Anoperineal Physiotherapy for Adult Anal Incontinence. Assessment of Incontinence Symptoms and Quality of Life.
Brief Title: ORALIA Trial Medical Treatment vs Anoperineal Physiotherapy for Adult Anal Incontinence.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 2006.429
Record Dates: First submitted 2006-10-12; First posted 2006-10-13 (Estimated); Last update posted 2013-09-19 (Estimated); Status verified 2013-09

CONDITIONS: Anal Incontinence
Keywords: Anal incontinence; Gastroenterology; Anoperineal physiotherapy; Randomized clinical trial
MeSH Terms: conditions — Encopresis

ARMS (2):
- standard medical treatment (Experimental): standard medical treatment
  Interventions: Behavioral: Standard medical treatment
- standard medical treatment + anoperineal physiotherapy (Experimental): standard medical treatment + anoperineal physiotherapy
  Interventions: Behavioral: standard medical treatment + anoperineal physiotherapy.

INTERVENTIONS:
Behavioral: standard medical treatment + anoperineal physiotherapy.
  Arms: standard medical treatment + anoperineal physiotherapy
Behavioral: Standard medical treatment
  Arms: standard medical treatment

SUMMARY:
The purpose of this study is to evaluate the impact of anoperineal physiotherapy in adjunction to standard medical treatment on symptoms and quality of life of adults with anal incontinence, in comparison with standard treatment alone.

A total of 443 patients will be randomized to 2 groups: standard care (medical treatment) alone or standard care associated with anoperineal physiotherapy. Outcome measures include the patient own view of the effectiveness of the treatment, the continence score, quality of life and psychological status. These outcomes are measured at the end of the 4 months treatment period.

Following this period, the non responders to standard medical treatment will be proposed to undergo a course of anoperineal physiotherapy and the non responders to anoperineal physiotherapy will be treated by transcutaneous electrical nerve stimulation (TENS). The outcomes will be measured at the end of the 4 months new treatment and again after 4 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 75
* Anal incontinence for more than six months.
* Signed informed consent
* Jorge and Wexner's anal incontinence score > or egal 5

Exclusion Criteria:

* Previous course of anoperineal physiotherapy within the past 6 months
* Anorectal or perineal surgery within the past 6 months.
* Indication for anoperineal surgery
* Vaginal delivery within the past 6 months
* Pregnancy
* Major neurological disease,
* Significant cognitive impairment, dementia or institutionalised.
* Active inflammatory bowel disease.
* Current treatment by sacral nerve neurostimulation.
* Cardiac pacemaker
* Skin damages preventing transcutaneous electrical nerve stimulation (TENS).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2006-10; Primary Completion 2011-06 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
The primary outcome variable is the patient's response to the question "How would you grade your symptom": major aggravation; aggravation, no changes, improvement and major improvement and rating of that change on an ordinal scale of -5 to +5. The p | during the treatment period

SECONDARY OUTCOMES:
Secondary outcomes include patient's symptoms questionnaire, continence score, quality of life questionnaire, stool diary and psychological status. These secondary outcomes are measured at the end of the 4 months treatment period and the end of follow-up | at the end of the 4 months treatment period and the end of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: François MION, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Anne-Marie SCHOTT, Lyon, France